CLINICAL TRIAL: NCT01715935
Title: A Comparison of Blood and Tissue Biomarkers Before and After Nephrectomy in the First-line Setting With Everolimus in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Biomarkers Before and After Nephrectomy of Locally Advanced or Metastatic Renal Cell Carcinoma Treated With Everolimus
Acronym: NEORAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-000882-11
Record Dates: First submitted 2012-09-12; First posted 2012-10-29 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-02

CONDITIONS: Clear-cell Renal Carcinoma; Clear-cell Metastatic Renal Cell Carcinoma
Keywords: Clear cells renal carcinoma; everolimus; neo-adjuvant treatment
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus (Experimental): everolimus, 10 mg PO daily. Before nephrectomy: 6 continuous weeks of treatment and one week of rest After nephrectomy: 4 weeks courses (for metastatic patients only)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — everolimus, 10 mg PO daily. Before nephrectomy: 6 continuous weeks of treatment and one week of rest After nephrectomy: 4 weeks courses (for metastatic patients only)
  Other Names: AFINITOR

SUMMARY:
Disease and Stage: Metastatic and locally advanced clear cell renal carcinoma

An open-label, exploratory, single-arm, multicenter trial.

Everolimus will be administered orally, once daily, for 6 weeks followed by a 1-week rest period prior to nephrectomy.

Two to four weeks after surgery, everolimus will be reintroduced only for metastatic patients until disease progression, unacceptable toxicity, withdrawal of patient consent, or other stopping rules are met.

DETAILED DESCRIPTION:
An open-label, exploratory, single-arm, multicenter trial. Treatment with everolimus will be initiated once patients have undergone baseline screening and provided their written informed consent.

Everolimus will be administered orally, once daily, for 6 weeks followed by a 1-week rest period prior to surgery. The starting dose will be 10 mg daily with provision for dose reduction based on tolerability.

Radical nephrectomy will be performed at the end of week 7. For metastatic patients, two to four weeks after surgery, everolimus will be reintroduced. Treatment will be continued until disease progression, unacceptable toxicity, withdrawal of patient consent, or other stopping rules are met.

Patients with locally advanced renal carcinoma will stop drug intake before nephrectomy.

Resumption of everolimus may be postponed in cases of a delay in wound healing or surgical complications.

After treatment discontinuation and the last treatment visit (28-days after the last dose), patients will be followed up in order to collect data on the onset of progression and survival. In metastatic patients discontinuing treatment for reasons other than disease progression, tumor assessment will continue every 3 months, until disease progression or initiation of other anticancer therapy for up to one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Advanced RCC or a resectable renal tumor and at least one measurable inoperable metastasis (at least 1 cm), in whom anti-angiogenic therapy is indicated
* Patients without target lesions, with bone metastasis
* Histologically confirmed clear cells RCC and possibility of adequate tumor sampling prior to treatment
* No prior systemic treatment for RCC
* Male or female, at least 18 years
* PS ECOG 0-1
* Life expectancy at least 3 months
* Adequate organ function with the following criteria:

  * Total serum bilirubin equal or less than 2 x ULN (Gilbert's disease exempted)
  * Serum transaminases and alkaline phosphatases equal or less than 2.5 x ULN, or in case of liver or bone metastasis equal or less than 5x ULN
  * Serum creatinine equal or less than 2 x ULN, creatinine clearance at least 50 ml/min
  * Absolute neutrophil count (ANC) at least 1500/mm3
  * Platelets at least 100,000/mm3
  * Hemoglobin at least 10.0 g/dL
  * INR equal or less than 1.7 or prothrombin time (PT) equal or less than 6 sec
  * Blood glucose less than 1.5x ULN
  * Fasting cholesterol equal or less than 5 mmol/L, triglycerides equal or less than 200 mg/dl,
* Negative pregnancy test within 7 days prior to enrollment
* Signed and dated IRB/ICE-approved informed consent form
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Patient covered by the national health system

Exclusion Criteria:

* Previous nephrectomy
* Histology: any histologic type different than ccRCC
* Treatment in a clinical trial in the last 30 days
* Previous treatment with everolimus or other mTOR-inhibitors and anti-angiogenic drugs
* Any of the following within 12 months prior to treatment initiation: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, ischemic or hemorrhagic stroke including transient ischemic attack, abnormal lung function.
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical treatment
* Abnormal ECG (Clinically significant)
* Treatment with vitamin K antagonists. Ongoing treatment with therapeutic doses of coumarin derivative anticoagulants (e.g. warfarin) or treatment within the 2 weeks before the first day of everolimus administration. Prophylaxis with low dose warfarin for deep vein thrombosis is permitted (up to 2 mg/day). Low molecular weight heparin is allowed.
* Brain metastasis. (Brain scan or MRI is mandatory). Note: Previous treated brain metastasis (surgery ± radiotherapy, radiotherapy, radiosurgery or gammaknife) and satisfying the following three criteria are allowed:

  * Asymptomatic;
  * No evidence of any active brain metastasis 3 months prior inclusion;
  * No necessity of corticoid or antiepileptic treatment.
* Pregnancy or breastfeeding.
* Any second malignancy within the last 3 years with the exception of basal cell carcinoma, in situ cervical cancer and pT1/a bladder cancer with no evidence of recurrent disease for 12 months.
* Clinically significant gastrointestinal abnormalities including but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel that could affect the absorption of the study drug
  * Active peptic ulcer disease
  * Inflammatory bowel disease
  * Ulcerative colitis or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
  * Hepatitis B/C
* Hypersensitivity to everolimus or any excipient of everolimus.
* Any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Objective clinical benefit | After 6 weeks of treatment
  Objective clinical benefit is defined as complete response, partial response or stable disease according to RECIST criteria version 1.1

SECONDARY OUTCOMES:
Progression Free Survival | up to 1 year
Overall survival | up to 2 years
Safety and tolerability | Participants will be followed all along the treatment period, an expected average of 15 months
  Toxicity will be classify according to NCI-CTC criteria Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Oudard, MD, PhD, Principal Investigator — Hôpital Européen Georges Pompidou, Paris (France)
Locations (10):
- France (10):
  - CHRU Besançon, Besançon
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hôpital Saint Eloi - CHU Montpellier, Montpellier
  - Fôpital d'Instruction des Amées du Val de Grâce, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou - Service d'oncologie médicale, Paris
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No